CLINICAL TRIAL: NCT02365428
Title: Pregnancy and Physical Activity: Text-message Referral to Evidence-based Websites
Brief Title: Evidence-based Websites to Increase Physical Activity for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1307009388
Record Dates: First submitted 2014-12-30; First posted 2015-02-19 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2015-02

CONDITIONS: Pregnancy
Keywords: Maternal welfare

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control: Group 1 (Experimental): The control group will receive three standard Text4Baby messages per week at noon on Mondays, Wednesdays, and Fridays.
  Interventions: Behavioral: Physical activity text messages
- Group 2 (Experimental): Intervention group 1 will receive two physical activity messages and one standard Text4Baby message each week at noon on Mondays, Wednesdays, and Fridays.
  Interventions: Behavioral: Physical activity text messages
- Group 3 (Experimental): Intervention group 2 will receive six physical activity messages and one standard Text4Baby message per week at a random time per day.
  Interventions: Behavioral: Physical activity text messages
- Group 4 (Experimental): Intervention group 3 will receive six physical activity messages and one standard Text4Baby message per week at a time of the participant's choice per day.
  Interventions: Behavioral: Physical activity text messages

INTERVENTIONS:
Behavioral: Physical activity text messages

SUMMARY:
Fewer pregnant women achieve recommendations for physical activity (PA) (30 minutes of moderate PA 5 days of the week) as compared to non-pregnant women (15.8% to 26.1% respectively), and PA participation declines as pregnancy progresses. The benefits of PA during pregnancy are abundant to both the mother (e.g., reduced weight gain, lower risk of gestational diabetes) and the fetus (e.g., decreased fat mass, improved stress tolerance). Pregnancy represents a significant time in a woman's life in which she may be motivated to change her health behaviors due to concerns for the healthy development of the fetus and a quick return to pre-pregnancy weight. Hence, pregnancy represents a critical time to support women in PA participation.

In our previous research, 94% of pregnant and postpartum women of varying socioeconomic statuses reported using the Internet for pregnancy and PA information. Despite some women increasing their PA participation as a result, most did not know if a website was reputable or reliable (i.e. evidence-based). Studies have reported that most online health information is unregulated and inaccurate. Further, women often receive inadequate PA information from physicians who are constrained by time and lack of knowledge about PA. Therefore, directing pregnant women to evidence-based websites via text messaging may provide a feasible approach to improve PA participation. PA participation in pregnant women is an ongoing challenge that warrants testing of innovative solutions.

The purpose of this study is to determine the feasibility of using mobile phone text messaging to refer pregnant women to evidence-based websites for PA information to increase PA levels.

DETAILED DESCRIPTION:
During Phase 1, the investigators will identify and test evidence-based websites and text messages with our target population.

First the investigators will conduct interviews with pregnant women who meet physical activity recommendations (n=15-20) (30 minutes of moderate intensity activity at least five days per week) to ask them about what helps them to be active during their pregnancy. Using the information gathered from these interviews and the literature the investigators will develop text messages and 200-300 word mobile (i.e., cell phone, tablet computer) websites. The mobile websites will include content from evidence-based websites, but will be adapted for the mobile platform to enhance the user interface and readability of the websites. The goal of the mobile websites is to allow women to access the websites by clicking on the link in each text message. Once developed, the first draft of evidence-based websites and text messages will be tested with interviews (pregnant women n=12, physician n=12, nurses/staff n=12) prior to their use. All phase one participants will be recruited through word of mouth, community nurse clinics and physician offices. Consultant Link will direct efforts to recruit participants from community nurse clinics. Dr. Coonrod, Dr. Huls and Ms. Braescu will direct efforts to recruit participants from physician offices. The purpose of the interviews are to determine the feasibility (perceived acceptability and demand) and the appropriateness (culturally and linguistically) of the material. A moderator and note-taker (student researchers) trained by the PI (Huberty) and Co-I (Hekler) will conduct interviews. All participants will receive $25 for their participation. The interviews will inform the second draft of evidence-based websites and text messages, which will be used to implement the intervention. An amendment that requests the approval of the text messages and websites will be submitted after the completion of Phase 1 and prior to the commencement of Phase 2.

Addition to Phase 2 - The investigators will conduct a survey to determine the appropriate dose (frequency and intensity) of physical activity text messages for Phase 2. The investigators will use this information to determine how often during the pregnancy (e.g., daily, weekly) and when during the pregnancy (e.g., first, second, third trimester, or throughout) that text messages with physical activity information are necessary to help women participate in physical activity during their pregnancy. The survey is approximately 45 questions in length and takes about 5 minutes to complete. Pregnant women will be recruited using word of mouth, fliers in places where pregnant women may be present (e.g., baby stores, maternity stores, community nurse clinics and physician offices,), email list servs (e.g. partnerships with Text 4 Baby and foundations related to pregnancy), and social media (e.g., Facebook, twitter). The investigators will recruit 200 women to complete the survey.

During Phase 2, the investigators will recruit women (n=75-100) to receive text messages referring them to evidence-based websites for PA information. Flyers will be available in physicians' clinics for posting and/or handout to women attending their first visit (8-16 weeks gestation). The PI will present the study information to physicians, nurses, and staff at all physicians' sites; however, physicians, nurses, and staff will only participate in passive recruitment methods via the study flyer. Participants will also be recruited nationally using social media (i.e., Facebook, Twitter) and word of mouth (i.e., emails). Interested participants will contact the research team (contact information on the flyer) to learn more about the study and complete the eligibility questionnaire. After completing the eligibility questionnaire (see attached), participants will be contacted via email to set up a time to complete an intake appointment. Intake appointments (to review and sign the informed consent form, discuss the study in more detail) with participants will take place over the phone. The participants' informed consent and baseline questionnaires must be received before they will be eligible to begin the intervention.

Participants will be assigned to a control group (n=25) or one of two intervention groups (n=50). The control group will receive three standard Text4Baby messages per week. Intervention group 1 will receive two physical activity messages and one standard Text4Baby message each week. Intervention group 2 will receive six physical activity messages and one standard Text4Baby message per week. The physical activity text message will refer the participant to an evidence-based (HON Code certified) website that includes PA information relative to the time in their pregnancy. Text messages will be pulled from a list of 150 possible text messages. The text messages and websites will provide educational information about PA and its health benefits, but women will not be given a prescribed PA program to follow as a part of this study. Therefore, a doctor's note approving women's participation in this study is not necessary.

All Phase 2 participants will be objectively measured for physical activity using the Fitbit activity monitor. The device will be mailed to women after completing the intake appointment and returning the informed consent and baseline questionnaires. The women will wear the device for 24 hours daily and will be asked to sync their device to their computer in order to send researchers their physical activity feedback. All Fitbit monitors will be identified only by a participant code to maintain the confidentiality of data when participants send their data via wireless internet and when researchers receive the data. Women will also be asked to complete short satisfaction surveys about some of the text messages. Fifteen women will receive the satisfaction surveys once per week, and 60 women will receive the surveys twice per month. The satisfaction survey is included with this application.

After the intervention, Phase 2 participants will be invited to participate in a voluntary interview to further examine the feasibility of the intervention. Areas of focus will include: acceptability (satisfaction, intention to use, perceived appropriateness), demand (actual use, intention to use), and implementation (factors affecting ease or difficulty) of using text messaging for referral to evidence-based websites for PA information. The interview can be conducted in person or over the phone. Participants who complete the intervention will be able to retain the FitBit device for their personal use.

Following the interview, participants will be invited to participate in Phase 3 of the study (Part 2) (new consent form).

During Phase 3 (Part 2), the information collected on the Fitbit physical activity monitor and synced with the user ID will be recorded during the mother's first year post-partum (from time of birth until the child's first birthday) just as it was during the pregnancy. The investigators will also send a survey, via a Qualtrics link, to complete every three months (4 times total) during this first year post-partum. The survey will ask questions related to mental health (i.e., stress, anxiety), physical health (i.e., weight, physical activity participation), and psychosocial characteristics (i.e., mood, support).

All Phase 3 (Part 2) participants will complete a new informed consent document in which they are aware that the investigators will continue to monitor their physical activity (without text messages) and will complete 4 surveys.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

* physician, nurse/staff, or pregnant patient at one of the participating physician sites
* able to speak English
* willingness to participate in one 1-hour interview
* 18 years of age or older.

Inclusion Criteria (Part 2 of Phase 1)

* pregnant or has been pregnant
* able to speak English
* willingness to participate in the 5 minute survey
* 18 years of age or older.

Inclusion Criteria (Phase 2)

* 8-20 weeks gestation
* 18 years of age or older
* own a smartphone with text message capability
* regular access to a computer
* ability to speak/read/understand English
* resident of the United States
* willingness to provide the research team with cell phone number to receive text messages
* not currently meeting physical activity guidelines of 30 minutes of moderate physical activity 5 days of the week.

Exclusion Criteria:

* pregnant women who are high risk as defined by the absolute and relative contraindications of exercise outlined in The American Congress of Obstetricians and Gynecologists' Position Statement on Exercise During the Pregnancy and Postpartum Period
* women who have physical limitations to physical activity
* women whose doctors instruct them NOT to be physically active during pregnancy and
* women who are currently meeting the physical activity recommendations of 30 minutes of moderate physical activity 5 days of the week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of Minutes Spent Doing Physical Activity Measured via a Physical Activity Monitor (FitBit) | 20 to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, Ph.D., Principal Investigator — Arizona State University